CLINICAL TRIAL: NCT01915758
Title: A Single-Center, Evaluator-Blinded, Randomized, Placebo-Controlled, Phase 1 Clinical Trial Evaluating the Photoallergic Potential of Topically Applied Clindamycin Phosphate 1.0% and Tretinoin 0.025% (CT Gel) in Healthy Volunteers
Brief Title: W0265-104: A Single-Center, Evaluator-Blinded, Randomized, Placebo-Controlled, Phase 1 Clinical Trial Evaluating the Photoallergic Potential of Topically Applied Clindamycin Phosphate 1.0% and Tretinoin 0.025% (CT Gel) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 114730
Record Dates: First submitted 2012-10-11; First posted 2013-08-05 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Gels

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- occlusive patch 200 uL of clindamycin1%/tretinoin0.025% Gel (Experimental): occlusive patch 200 uL of clindamycin1%/tretinoin0.025% Gel
  Interventions: Drug: clindamycin1%/tretinoin 0.025% gel
- occlusive patch 200uL of vehicle gel (Placebo Comparator): occlusive patch 200uL of vehicle gel
  Interventions: Drug: vehicle gel

INTERVENTIONS:
Drug: clindamycin1%/tretinoin 0.025% gel — clindamycin1%/tretinoin 0.025% gel
  Arms: occlusive patch 200 uL of clindamycin1%/tretinoin0.025% Gel
Drug: vehicle gel — vehicle gel
  Arms: occlusive patch 200uL of vehicle gel

SUMMARY:
This was a single-center, evaluator-blinded, randomized, placebo (vehicle) -controlled phase I study to evaluate the photoallergic potential of Clindamycin-Tretinoin Gel. The design consisted of the following periods: screening, induction, rest, challenge, and rechallenge (if indicated). Induction visit 1 was to occur within 5 days of screening visit 2. The study expected to enroll approximately 62 healthy adult volunteers. Subjects were to receive repeated 24-hour study patch applications; after patch removal, the sites were irradiated with ultraviolet B light (UVB) and visible light (VIS) during the induction period (consisting of 6 consecutive induction phases), and ultraviolet A light (UVA)/ UVB and VIS during the challenge and rechallenge periods. Each application site was observed approximately 1, 24, 48, and 72 hours later for signs of inflammation.

DETAILED DESCRIPTION:
This was a single-center, evaluator-blinded, randomized, placebo (vehicle) -controlled phase I study to evaluate the photoallergic potential of Clindamycin-Tretinoin Gel. The design consisted of the following periods: screening, induction, rest, challenge, and rechallenge (if indicated). Induction visit 1 was to occur within 5 days of screening visit 2. The study expected to enroll approximately 62 healthy adult volunteers. Subjects were to receive repeated 24-hour study patch applications; after patch removal, the sites were irradiated with ultraviolet B light (UVB) and visible light (VIS) during the induction period (consisting of 6 consecutive induction phases), and ultraviolet A light (UVA)/ UVB and VIS during the challenge and rechallenge periods. Each application site was observed approximately 1, 24, 48, and 72 hours later for signs of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* The capability of understanding and providing signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol-specific procedures were performed.
* Male or female subjects aged from 18 to 65 years, inclusive, at time of consent.
* The ability to complete the study and to comply with study instructions.
* Possessed Fitzpatrick skin type I (always burns easily; never tans), II (always burns easily; tans minimally), or III (burns moderately, tans gradually) that would not interfere with the reading of any skin responses. Determination of skin types was based on sunburn and tanning histories, as well as subjects' opinions of their responses to the first 30 to 45 minutes of sun exposure.
* Sexually active females of childbearing potential who agreed to use a medically acceptable method of contraception while receiving protocol-assigned product. A woman of childbearing potential was defined as one who was biologically capable of becoming pregnant, including perimenopausal women who were less than 2 years from their last menses. Acceptable contraceptive methods included the following:
* Hormonal contraception, including oral, injectable, or implantable methods started at least 2 months prior to screening. If hormonal contraception was started less than 2 months prior to screening, then a form of non-hormonal contraception was to have been added until the third continuous month of hormonal contraception was completed.
* Two forms of non-hormonal contraception, including intrauterine devices or properly used barrier methods (eg, male or female condoms, diaphragm, or cervical cap). Subjects with surgical sterilization, including tubal ligation or partner's vasectomy, were to have used a form of non-hormonal contraception. A barrier method or sterilization plus spermatocide were acceptable.
* Women who were not currently sexually active or lactating agreed to use a medically accepted method of contraception is she became sexually active while participating in the study.

Exclusion Criteria:

* Currently diagnosed with cancer or had a previous history of cancer, including skin cancer, or severe photodamaged skin. Severe photodamaged skin was characterized by yellow-gray color, wrinkles with no visible normal skin, and prior skin malignancies.
* Female subjects who were pregnant, attempting to become pregnant, or breast feeding.
* Received any investigational drug within 4 weeks of study day 1 or who were scheduled to receive an investigational drug other than the study product during the study.
* Used contraindicated prescription drugs within 4 weeks or 5 half-lives, whichever was longer, of first dose of study product, unless agreed as not clinically relevant by the principal investigator and the project physician.
* Participated in a previous study of the same study product.
* Current use of any medication which, in the opinion of the investigator, may have affected the evaluation of the study product or placed the subject at undue risk.
* Suffered from any disease or condition which, in the opinion of the investigator, may have affected the evaluation of the study product or placed the subject at undue risk.
* Any major illness within 30 days before the screening examination.
* Considered immunocompromised or using immunosuppressant drugs.
* Clinically relevant history of or current evidence of abuse of alcohol or other drugs.
* History of known or suspected intolerance to any of the ingredients of the study products (ie, test and comparator products), to the hypoallergenic tape, or to the cotton patches.
* Clinically relevant history or presence of respiratory (including chronic asthma requiring repetitive drug interventions), gastrointestinal, renal, hepatic, hematological, lymphatic, immunological, dermatological, or connective tissue diseases or disorders.
* Considered unable or unlikely to attend the necessary visits.
* History of severe reactions from exposure to sunlight, including previous experience with photoallergy, solar urticaria, polymorphous light eruptions, or other photo-exacerbated systemic diseases.
* Current use or expected use of photosensitizing medications (over-the counter and prescription), herbal supplements, or any use of a known photosensitizing material.
* Clinically significant skin diseases contraindicating participation or interfering with test site evaluations, including psoriasis, eczema, atopic dermatitis, acne, dyplastic nevi, or other skin pathologies.
* Investigator inability to evaluate the skin in and around the potential test sites due to sunburns, unevenness in skin tones, tattoos, scars, excessive hair, freckles, birthmarks, moles, or other skin abnormalities.
* Used topical medications (eg, corticosteroids or immunosuppressives) on potential test sites within the last 7 days prior to screening visit 1.
* Currently receiving allergy injections, or due to receive an injection, within 7 days prior to screening visit 1, or expected to begin injections during study participation.
* Used antihistamines or prescription anti-inflammatory drugs within 72 hours of the day 1 visit. Permitted exceptions were acetaminophen at recommended doses and aspirin at doses of less than 81 mg/day.
* Participated in any patch test study for irritation or sensitization or any test involving ultraviolet exposures within the last 4 weeks.
* Employees of the CRO or sponsor involved in the study, or an immediate family member (partner, offspring, parents, siblings, or sibling's offspring) of an employee involved in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-11-21 (Actual); Primary Completion 2009-02-20 (Actual); Study Completion 2009-02-20 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be inflammatory response or superficial effect at challenge period. Inflammatory responses (erythema and local skin reactions) or superficial effects (if observed) will be scored according to the grading scales. | Day 44 - 65
  In cases where the patch area is larger than the irradiated area, only the irradiated areas will be scored unless reactions outside the irradiated area exhibit unusual responses. Scores represent the presence of clinically significant effects on at least 25% of the test site. Questionable, barely perceptible, or minimal reactions involving less than 25% of the test site will not be considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- See also: Results for study 114730 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/114730?search=study&search_terms=114730#rs